CLINICAL TRIAL: NCT01660425
Title: Enhancement of Psychosocial Functioning, Quality of Life, Satisfaction With Medication and Medication Compliance of Methylphenidate Treatment by Psychosocial Intervention and Support
Brief Title: Enhancement of Methylphenidate Treatment by Psychosocial Intervention and Support
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Cologne (Other)
Collaborators: Shire (Industry)
Responsible Party: Principal Investigator, Manfred Doepfner, Leading psychologist at the Department of Childhood and Adolescence Psychiatry, University of Cologne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADHD-TEAM-02; 2486738 (Other Grant/Funding Number: Shire pharmaceutical development limited)
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Attention Deficit-/Hyperactivity Disorder
Keywords: Attention deficit-/hyperactivity disorder; parenting enhancement training; guided self-help; methylphenidate
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Psychosocial Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- treatment as usual with MPH (No Intervention): In the first twelve months of intervention the children receive treatment as usual with MPH and do not get any further intervention. Afterwards, the families get the opportunity to take part in the program which is then conducted for a duration of four months. Measurements are performed at the beginning of the program, after six moths, after 12 months and additionally after 16 months.
- Psychosocial intervention (Active Comparator): Parenting Enhancement Training as a form of psychosocial intervention is a guided program. Parents get the opportunity to discuss written information with a therapist in 20 minutes telephone calls. 14 telephone calls are offered. The whole intervention lasts for a period of one year. Booklets are mailed via post within the first 4 months. First 9 telephone calls are also within the first 4 months, usually every two weeks. Telephone calls 10 and 11 are within 5th or 6th month, telephone calls 12 to 14 are within 7th to 12th month with a two monthly time period in between.
  Interventions: Behavioral: Enhancement with psychosocial intervention

INTERVENTIONS:
Behavioral: Enhancement with psychosocial intervention
  Arms: Psychosocial intervention

SUMMARY:
The main purpose of this study is to evaluate the effectiveness of a parenting enhancement training (PET) for parents with children diagnosed with Attention Deficit-/Hyperactivity Disorder (ADHD) who are already medicated with methylphenidate.

DETAILED DESCRIPTION:
The main purpose of this study is to evaluate the effectiveness of a parenting enhancement training (PET) for parents with children diagnosed with Attention Deficit-/Hyperactivity Disorder (ADHD) already medicated with methylphenidate (MPH). This particular PET was developed at the Department of Child and Adolescent Psychiatry and Psychotherapy at the University of Cologne and has already been evaluated in several studies. MPH treatment has been proven to be efficacious in the reduction of ADHD symptoms. However, despite optimal titration a substantial percentage of children still suffer from residual symptoms and impairment in psychosocial functioning. Therefore, there is still room for improvement in satisfaction with medication. Moreover, a substantial rate of patients with good treatment effects fails to comply with medication during the course of treatment. This parenting enhancement training (PET) mainly conducted via written materials and telephone support will be introduced in patients already treated with MPH. Effects are expected on symptoms of ADHD as well as on comorbid oppositional symptoms. Further outcome parameters are satisfaction with medication and medication compliance of MPH treatment, psychosocial functioning as well as parenting skills. Parenting skills are a main focus of the PET and ADHD symptoms shall be improved through improving parenting skills. Besides focusing on symptoms, recent research often focuses on improvement of quality of life and impairment in psychosocial functioning (e. g. family, school, leisure time) as well. Not only suffer patients from the main symptoms. Many patients suffer as well from the symptoms' consequences, which is often an overall impairment. Satisfaction with medication and medication compliance are fundamental conditions for the success of a long term medical therapy. However, many studies show a lack of compliance.

ELIGIBILITY:
Inclusion Criteria:

* The child attends school and is aged 6 to 12
* Primary diagnosis of ADHD
* Medication with methylphenidate in stable doses for at least two months
* Currently, no change of medication is planned
* The parents are motivated to participate in the parenting enhancement training
* The parents have a command of written and spoken German
* Psychosocial impairment measured with WFIRS-P

Exclusion criteria:

- the family takes presumably part in psychotherapy with an intensive parenting training component during the duration of the intervention

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2012-05; Primary Completion 2014-12 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Change in Weiss Functional Impairment Rating Scale (WFIRS-P), parent rating | baseline, six months, 12 months; 16 months (control group)
  The WFIRS-P is used for the assessment of psychosocial functioning of children diagnosed with ADHD.

SECONDARY OUTCOMES:
Change in Symptom Checklist for Attention Deficit/Hyperactivity Disorder (FBB-ADHS), parent rating | baseline, six months, 12 months; 16 months (control group)
  The FBB-ADHS is used to assess symptoms of ADHD according to DSM-IV and ICD-10 rated by a parent.
Change in Symptom Checklist for Oppositional Defiant and Conduct Disorder (FBB-SSV), parent rating | baseline, six months, 12 months; 16 months (control group)
  The Symptom Checklist for Oppositional Defiant and Conduct Disorder (FBB-SSV) is used to assess symptoms of ODD and some of the symptoms of Conduct Disorders according to ICD-10 and DSM-IV.
Change in Individual Problem Checklist (IPC), parent rating | baseline, six months, 12 months; 16 months
  The IPC assesses individual problems as defined together with the parents. It represents the individual problems which were aimed to reduce with the treatment.
Change in Satisfaction with Medication Scale (SAMS), parent rating | baseline, six months, 12 months; 16 months (control group)
  The SAMS is used to assess parents' satisfaction with the medication of their child as well as with the effects of medication.
Change in "Compliance Scale", parent rating | baseline, six months, 12 months; 16 months (control group)
  Newly developed parent questionnaire consisting of five items to assess the medication compliance of the patient
Questionnaire to assess adverse effects of medication, taken from the Day Profile of ADHD Symptoms (DAYAS) | baseline, six months, 12 months; 16 months (control group)
  Subscale of the Day Profile of ADHD Symptoms (DAYAS) which assesses in 11 items the most frequent side effects of ADHD medication

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Doepfner, PhD, Principal Investigator — University of Cologne
Locations (1):
- Department of Child and Adolescent Psychiatry and Psychotherapy at the University of Cologne, Cologne, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Dose C, Hautmann C, Buerger M, Schuermann S, Woitecki K, Doepfner M. Telephone-assisted self-help for parents of children with attention-deficit/hyperactivity disorder who have residual functional impairment despite methylphenidate treatment: a randomized controlled trial. J Child Psychol Psychiatry. 2017 Jun;58(6):682-690. doi: 10.1111/jcpp.12661. Epub 2016 Nov 23. PMID 27878809